CLINICAL TRIAL: NCT07266948
Title: Evaluating the Impact of TRYPTYR on a Patient's Quality of Life and Ability to Perform Work
Brief Title: Impact of TRYPTYR on a Patient's Quality of Life and Ability to Perform Work
Acronym: TRYPTYR ADL
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Southern College of Optometry (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00006763-ADL
Record Dates: First submitted 2025-11-25; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Dry Eye; Eye Diseases; Eyes Dry Chronic
MeSH Terms: conditions — Dry Eye Syndromes; Eye Diseases

STUDY DESIGN:
Intervention Model Description: Qualifying participants will be given and instructed on appropriate dosage of using Acoltremon 0.003% TRYPTYR to determine i it alleviates the symptoms associated with Dry Eye Disease
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- TRYPTYR (Experimental): Participants who qualify for the study will be given TRYPTYR to determine if it is able to help alleviate symptoms associated with dry eye disease;
  Interventions: Drug: Acoltremon

INTERVENTIONS:
Drug: Acoltremon — Participants will be provided with Acoltremon or TRYPTYR to determine whether or not it is an effective medication to help alleviate symptoms associated with dry eye disease

SUMMARY:
This 1-month, 3-visit study will be conducted at the Southern College of Optometry (Memphis, TN), Kannarr Eye Care, LLC (Pittsburg, KS) and Complete Eye Care of Medina (Minneapolis, MN). Adults ≥18 years of age who have been diagnosed with DED for at least 6 months and who are currently symptomatic (Eye Dryness VAS Score ≥40) will be recruited. Subjects will have an abnormal Schirmer test of <10 mm/5 min. Subjects will also be required to score ≤70 on the IDEEL Quality of Life (QoL) Work domain to ensure that their DED symptoms are significantly impacting their ability to do work.9 Subjects will be required to have corrected distance visual acuity of 20/32 (0.2 logMAR) or better.

DETAILED DESCRIPTION:
Dry eye disease (DED) is a prevalent condition that commonly affects patients of working age in addition to the elderly.1-3 DED is a complex condition that results in ocular symptoms such as dryness and burning and signs such as decreased tear production (aqueous deficient DED) or increased tear evaporation (evaporative DED).4 Unfortunately, there is not a perfect correlation between DED signs and symptoms,5 which makes diagnosis and timely treatment challenging. With DED symptoms often being bothersome and there being a lack of universally effective treatment options,6 DED patients are significantly more likely to suffer from a decreased quality of life and a psychological condition such depression.7 Thus, the DED patient population would strongly benefit from new, innovative treatments that are based upon a novel mechanism.

Acoltremon 0.003% (TRYPTYR; Alcon Laboratories; Fort Worth, TX, USA) was recently approved by the US Food and Drug Administration (FDA) as the first transient receptor potential melastatin 8 (TRPM8) agonist for the treatment of DED.8 Acoltremon acts by activating TRPM8 receptors expressed on the neurons of the ophthalmic division of the trigeminal nerve, which is the nerve that innervates the cornea and eyelid.8 This drugs subsequently stimulates cold thermoreceptor to increase tear production. While acoltremon 0.003% has been significantly shown to improve tear production and symptoms as measured by the Symptom Assessment in Dry Eye (SANDE) at 14- and 28-days post-treatment, the community currently lacks data related to key measures of quality of life such as one's ability to work and perform daily tasks. Thus, the purpose of this study is to determine if acoltremon 0.003% can significantly improve the quality of life of DED suffers

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age.
* Have a history of DED for at least the past 6 months.
* Are currently using Restasis as directed by their eye care provider for ≥1 month.
* Participant intends to stop Restasis in the near future because and expressed dissatisfaction with effectiveness of Restasis in reducing dry eye symptoms..
* Are symptomatic as determined with the Eye Dryness visual analog scale (VAS) (Score ≥50), SPEED (≥7), and have an abnormal Schirmer test score [≥2 to <10 mm/5 min]) at Screening/Baseline.
* Have corrected distance visual acuity of 20/100 or better.
* Willing to discontinue contact lens wear throughout the study.

Exclusion Criteria:

* Have a systemic health condition that is known to alter tear film physiology (e.g., primary and secondary Sjögren's syndrome).
* Have a history of ocular surgery within the past 12 months.
* Have a history of severe ocular trauma, active ocular infection or inflammation that is not dry eye related.
* Punctal plugs in place for < 3 months and/or Lacrifill in place for > 5 months.
* Have ever used Accutane or are currently using ocular medications (must washout from all dry eye medications/treatments at least 1 week before entry, except for Restasis).
* Use of artificial tears within 2 hours prior to the baseline visit or during the study.
* Are pregnant or breast feeding.
* Have had a physical meibomian gland treatment withing 1 month of enrollment.
* Have a condition or be in a situation, which in the investigator's opinion, may put the participant at significant risk, may confound the results, or may significantly interfere with their study participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in IDEEL-QoL Work scores at 28 days. | 1 month
  the ideel quality of life questionnaire will be used to determine if there was an improvement in participant quality of life while using tryptyr

SECONDARY OUTCOMES:
Mean change from baseline in IDEEL-QoL Work scores at 14 days. | 14 days
  the ideel quality of life questionnaire will be used to determine if there was an improvement in participant quality of life while using tryptyr

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Kannar Eye Care, Pittsburg, Kansas
  - Complete Eye Care of Medina, Medina, Minnesota
  - The Southern College of Optometry, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided